CLINICAL TRIAL: NCT04832451
Title: Effects of Interpersonal Relational Role Analysis on Nursing Students' Depressive Symptoms and Coping Styles
Brief Title: Effects of Interpersonal Relational Role Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Yasemin Cekic, Research Assistant Dr., Ankara University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 56786525-050.04.04-6988
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Depressive Symptoms; Coping Skills
Keywords: coping styles; depressive symptoms; interpersonal relational role analysis; nursing students; stress
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: randomized controlled, pre-test-post-test control group design and follow-up test patterns
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The Beck Depression Inventory[BDI] (inclusion criteria) was applied face to face to the students who constituted the population (n=385). After the BDI scores were evaluated, the students who met the inclusion criteria were randomly assigned to the intervention and control groups.
  In a preliminary interview held with the intervention group (n=10), they were informed about the subject of the research, the duration and content of the implementation process, session rules, and that sessions would be audio-recorded. Informed consent forms were obtained from them, and pre-tests (BDI, Coping Styles Inventory[CSI]) were applied.
  A total of 21 90-minute Interpersonal Relational Role Analysis (IRRA) sessions (two sessions a week) were held with the intervention group.
  21 sessions of IRRA were applied to the intervention group, once the sessions were completed, post-tests (BDI, CSI) were applied. Three months later, a follow-up test (BDI, CSI) was applied to intervention group.
  Interventions: Behavioral: Interpersonal Relational Role Analysis
- Control Group (No Intervention): The students in the control group were informed about the research, informed consents were obtained from them, and pre-tests (Beck Depression Inventory, Coping Styles Inventory) were applied to them. No intervention was applied to the control group (n=10). Once the Interpersonal Relational Role Analysis sessions were completed, post-tests (Beck Depression Inventory, Coping Styles Inventory) were applied to the control group. Three months later, a follow-up test (Beck Depression Inventory, Coping Styles Inventory) was applied to control groups. After the follow-up test, the participants in the control group were referred to the psychological support unit of the university.

INTERVENTIONS:
Behavioral: Interpersonal Relational Role Analysis — Interpersonal Relational Role Analysis (IRRA) is a psychosocial group intervention that allows individuals to see the problems they experience in interpersonal relationships and interactions in the group environment and to be handled together with group members.
  Similar to Yalom's interactional group therapy model, IRRA sessions comprise warm up, the stages of setting the agenda, working, evaluating, and getting feedback from observers, which are based on the 'here and now' principle. IRRA helps to safely examine the roles in which group members are "stuck," in a group environment which is a small example of social life, and these roles are addressed in six steps.
  Arms: Intervention Group

SUMMARY:
Introduction: Interpersonal Relational Role Analysis (IRRA) is a psychosocial group intervention that allows individuals to see the problems they experience in interpersonal relationships and interactions in the group environment and to be handled together with group members.

Aim: The present study aims to investigate the effects of IRRA on nursing students' depressive symptoms and coping styles.

Method: This study was conducted with randomized controlled, pre-test-post-test control group design and follow-up test patterns. Students with depressive symptoms were randomly assigned to control (n=10) or intervention groups (n=10). Intervention group students received 21 weeks of IRRA intervention.

Results: It was determined that IRRA had a positive effect on nursing students' depressive symptoms and coping styles.

Discussion: This study is the first to evaluate the effects of IRRA on depressive symptoms and coping styles. Our study provides evidence on the effectiveness of IRRA in reducing the depressive symptoms of nursing students and in managing stress.

Implications for Practice: IRRA is a practical and useful intervention that mental health nurses can incorporate and use in their clinical practice while helping individuals to become aware of problems in relationships and roles that may impair their mental health.

DETAILED DESCRIPTION:
Aim and Design Aiming to investigate the effects of Interpersonal Relational Role Analysis (IRRA) on nursing students' depressive symptoms and coping styles, this study was conducted with randomized controlled, pre-test-post-test control group design and follow-up test patterns.

Research population and sample The study was conducted in the 2018-2019 academic year (November 2018 - April 2019). The research population comprised second-year nursing students studying at two different state universities in the 2018-2019 academic year (n=385). Since the researcher had an instructional relationship with the first-, third-, and fourth-year students, the study was performed with the second-year students. The number of people to be included in the groups was calculated in the G*Power (3.1.9.2) package program based on a research. As a result of the power analysis with an effect size of 0.7, a power of 80%, and an alpha level (probability of making a type I error) of 0.05, the sample size was calculated as a total of 16 students (8 in the intervention and 8 in the control group). Considering the possibility of drop-outs during the study, the research was conducted with a total of 20 students (10 in the intervention and 10 in the control group). Effective implementation of IRRA requires interaction among the group members; therefore, the intervention group was composed of students studying in the same class. To prevent interaction between the control group and the intervention group, the control group was composed of students studying at a different state university in the same city with the same education program. The students who met the inclusion criteria and agreed to participate in the study were assigned to the intervention and control groups with the Research Randomizer program. Randomization was performed by a researcher who was not included in the research. To make the study a single-blind study, students were not informed about the group to which they were assigned.

Inclusion/exclusion criteria Inclusion criteria were as follows: (a) being a nursing student at the university during the research (November 2018-April 2019), (b) not having any disability that would cause difficulties in filling in the data collection tools or during sessions, (c) scoring scores indicating mild to moderate depression from the Beck Depression Inventory, (d) agreeing to participate in the research, and (e) being over 18 years old. Exclusion criteria were as follows: (a) scoring scores indicating severe depression from the Beck Depression Inventory (severe depression requires psychopharmacological treatment).

Data Collection Tools Sociodemographic Characteristics Form This form, developed by the researchers, contains questions about students' sociodemographic characteristics such as age, gender, marital status, economic status, and parental educational status.

Beck Depression Inventory (BDI) The inventory consists of 21 self-report items that allow evaluating the severity of depressive symptoms rather than the diagnosis of depression. The total score obtained from the scale is evaluated, each item is scored between 0 and 3, and there are no reverse-scored items on the scale. 0-9 points indicate probably no depression, 10-16 points mild depression levels, 17-24 points moderate depression levels, and 25 and above points severe depression. The above-mentioned classification was used in this study. Cronbach's alpha reliability coefficient of the scale was calculated as 0.74.

Coping Styles Inventory (CSI) The scale has 30 items and five sub-dimensions rated on a four-point Likert-type scale. To calculate the score from the "seeking social support" sub-dimension, the first and ninth items are reversely scored. The scores of the sub-dimensions are calculated by dividing the total scores obtained from the items by the total number of items. High scores from the self-confident approach, optimistic approach, and seeking social support sub-dimensions indicate that effective methods are used to cope with stress whereas high scores from the helpless approach and submissive approach sub-dimensions indicate that ineffective methods are used to cope with stress. Cronbach's alpha reliability coefficient was calculated as 0.69 for the self-confident approach sub-dimension, 0.63 for the optimistic approach sub-dimension, 0.72 for the seeking social support sub-dimension, 0.67 for the helpless approach sub-dimension, and 0.68 for the submissive approach sub-dimension.

Implementation First, the BDI (inclusion criteria) was applied face to face to the students who constituted the population (n=385) (06-08 November 2018). After the BDI scores were evaluated, the students who met the inclusion criteria were randomly assigned to the intervention and control groups.

In a preliminary interview held with the 10 students in the intervention group, they were informed in a confidential manner about the subject of the research, the duration and content of the implementation process, what was expected from the participants, session rules, the place where the sessions would be held, and that sessions would be audio-recorded. Also, informed consent forms were obtained from them, and pre-tests (BDI, CSI) were applied (14 November 2018). Likewise, the students in the control group were informed about the research, informed consents were obtained from them, and pre-tests were applied to them (15 November 2018).

A total of 21 90-minute IRRA sessions (two sessions a week) were held with the 10 students in the intervention group between 16.11.2018 and 20.01.2019. The sessions were chaired by a group administrator (the researcher) and two observers (faculty members in the field of mental health nursing). The group administrator received IRRA training from faculty members who developed the IRRA model. Before the sessions, warm-up exercises were performed in order to develop a sense of trust and to increase rapport and interaction among the members. In the first session, an "acquaintance activity" was held, and the session rules, about which the participants were informed in the preliminary interview, were again presented for everyone's approval. In the following sessions, after the warm-up exercises, an agenda-setting round (a process devoted to setting the agenda) was carried out with the participation of each member. At this stage, each member was asked whether they experienced an important event they wanted to share with other members, and then each member summarized which IRRA step they were in and determined on which step they would work throughout that day's session. After this stage, the members who wanted to work in the group in that day's session worked on the IRRA steps. In each session, 45-50 minutes were allocated to examining the IRRA steps. During this time, participants were given opportunities to express themselves, and the IRRA steps of 2-3 members were discussed in each session, depending on the progress of the group members. Due to individual differences, some members made rapid progress through the IRRA steps, while it took others longer to complete the steps. At the end of each session, a 15-20 minute evaluation round was held with the participation of the observers. During the evaluation, the group administrator summarized what was discussed in the session. Participants were asked how they felt during the session, their negative feelings were studied, and it was ensured that no members left the session with negative feelings. The group administrator and observers gave empathic and positive feedback to each member due to their efforts to improve and change themselves. Similarities between the experiences and feelings of the participants were emphasized. The members thanked each other for confiding in each other. In the last session, a "separation activity" was held, where the members shared the positive aspects they discovered about each other, as well as their feelings and thoughts about the ending of the group.

While 21 sessions of IRRA were applied to the intervention group, no intervention was applied to the control group. Once the IRRA sessions were completed, post-tests (BDI, CSI) were applied to the intervention and control groups (January 21-24, 2019). Three months later (April 2019), a follow-up test (BDI, CSI) was applied to both groups. After the follow-up test, the participants in the control group were referred to the psychological support unit of the university.

Data Analysis Data were analysed using the Statistical Package for Social Sciences 22.0. In the evaluation of the data, the Kolmogorov-Smirnov test was applied to determine whether the data had a normal distribution or not, regarding the steepness and skewness. As a result of the analysis, it was found out that the significance value of the Kolmogorov-Smirnov test was higher than 0.05, the steepness and skewness values were between the range of -1 and +1, and the data had a normal distribution. The independent samples t test and chi-square test were used to examine the homogeneity of participant characteristics and outcome variables between the intervention and control group at baseline.

The versatile variance analysis was performed for the comparison of the group, time, and group×time interaction among means of BDI and CSI subscale score in the intervention and control groups. To compare the mean scores among the groups one-way variance analysis in repeated measurements was used, and "the Bonferroni-adjusted t test for dependent samples" was used to compare the measurements.

Ethical approval This study was approved by a research ethics committee (56786525-050.04.04-6988). Written and verbal consent was obtained from the students who agreed to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* being a nursing student at the university during the research (November 2018-April 2019),
* not having any disability that would cause difficulties in filling in the data collection tools or during sessions,
* scoring scores indicating mild to moderate depression from the Beck Depression Inventory,
* agreeing to participate in the research,
* being over 18 years old.

Exclusion Criteria:

* scoring scores indicating severe depression from the Beck Depression Inventory (severe depression requires psychopharmacological treatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory | 5 months
  The Turkish validity and reliability study of the inventory, which was developed by Beck et al. (1961), was conducted by Hisli (1989). The inventory consists of 21 self-report items that allow evaluating the severity of depressive symptoms rather than the diagnosis of depression. The total score obtained from the scale is evaluated, each item is scored between 0 and 3, and there are no reverse-scored items on the scale. 0-9 points indicate probably no depression, 10-16 points mild depression levels, 17-24 points moderate depression levels, and 25 and above points severe depression. The above-mentioned classification was used in this study. Cronbach's alpha reliability coefficient of the scale was calculated as 0.74 (Hisli, 1989).

SECONDARY OUTCOMES:
Coping Styles Inventory | 5 months
  The Turkish validity and reliability study of the scale, which was developed by Folkman and Lazarus (1980) to determine the ways to cope with stressful situations, was conducted by Sahin and Durak (1995). The scale has 30 items and five sub-dimensions rated on a four-point Likert-type scale. To calculate the score from the "seeking social support" sub-dimension, the first and ninth items are reversely scored. The scores of the sub-dimensions are calculated by dividing the total scores obtained from the items by the total number of items. Cronbach's alpha reliability coefficient was calculated as 0.69 for the self-confident approach sub-dimension, 0.63 for the optimistic approach sub-dimension, 0.72 for the seeking social support sub-dimension, 0.67 for the helpless approach sub-dimension, and 0.68 for the submissive approach sub-dimension (Sahin & Durak, 1995).

CONTACTS AND LOCATIONS:
Overall Officials: Gülsüm ANÇEL, PhD, Study Director — Ankara University
Locations (1):
- Ankara University Faculty of Nursing, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No